CLINICAL TRIAL: NCT03741088
Title: Multi-center, Open-labeled, Non-randomized Study to Evaluate the Acute Technical Performance and Safety Profile of the VORTX Rx® for Ablation of Primary and Metastatic Liver Tumors (Theresa Study)
Brief Title: Study to Evaluate VORTX Rx (Theresa)
Acronym: Theresa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HistoSonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 03.CP.0.3
Record Dates: First submitted 2018-07-19; First posted 2018-11-14 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Carcinoma, Hepatocellular; Liver Metastases
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- VORTX Rx treatment (Experimental): Focused ultrasound ablation of liver tumors.
  Interventions: Device: VORTX Rx treatment

INTERVENTIONS:
Device: VORTX Rx treatment — Cavitation-based cellular destruction using focused ultrasound

SUMMARY:
Multi-center, Open-labeled, Non-randomized Study to Evaluate the Acute Technical Performance and Safety Profile of the VORTX Rx® for Ablation of Primary and Metastatic Liver Tumors

DETAILED DESCRIPTION:
The study will assess the technical performance of the VORTX Rx device to deliver acoustic energy for cavitation-based cellular destruction. The planned duration of a single target tumor will be 60 minutes or less in a single session and adjusted intra-procedurally as necessary per investigator discretion. Subjects in this study must have an adequate acoustic window in the abdominal space in order to be eligible for enrollment. All patients who undergo ablation with the investigation device will be treated in a hospital environment under general anesthesia not to exceed four hours.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before any study procedure is performed.
* Subjects of both sexes aged 18 years or older.
* Patients diagnosed with liver cancer, including HCC or liver metastases from breast, pancreas and/or colorectal cancers. If biopsy is required, there will be a minimum of 2-week period after biopsy and before the ablation.
* HCC patients must meet the United Network for Organ Sharing and Organ Procurement and Transplantation Network (UNOS-OPTN) class 5 criteria for HCC (52).
* Liver metastases patients must meet minimum criteria of liver biopsy and/or tissue diagnosis of primary tumor or metastatic tumor with new or growing liver tumors radiologically consistent with metastases.
* Patients with liver cancer not candidates for surgical resection and/or not suitable for other locoregional treatments or patients who have not responded to or relapsed from conventional therapies.
* Previous treatment with chemotherapy and/or radiotherapy is permitted provided that these treatments have been discontinued more than 2 weeks before the ablation and whenever patients have recovered from any related toxicity (53).
* Previous treatment with immunotherapies is permitted provided that these therapies have been discontinued at least 4 weeks before the ablation and whenever patients have recovered from any related toxicity.
* Previous ablation/surgery on other tumors different from those that will be targeted with the VORTX Rx® is allowed whenever a minimum of 2 weeks has elapsed since the prior procedure(s).
* Tumor to be targeted for ablation will be clearly separated from other tumors or other critical areas (i.e. located in different segments of the liver) and located in segment 2, 3, 4, 5 or 6.
* Largest diameter of targeted tumor ≤3 cm.
* Tumor that will be targeted at a depth <10 cm from the skin surface.
* Must have an adequate acoustic window in the abdominal space to be able to visualize targeted tumor using ultrasound imaging; also must be able to visualize targeted tumor using MRI with optional CT imaging at investigator discretion.
* Patients who can undergo general anesthesia.
* Liver function score of Child-Pugh A or Child-Pugh B.
* ECOG PS 0, 1 or 2 at screening.
* Adequate liver function (ALT and AST < 2.5 x upper limit of normal [ULN]), renal function (serum creatinine <2 ULN and/or bilirubin <2.5 UNL) and hematologic function (neutrophil count > 1.0 x 109/L and platelet > 50 x 109/L).
* An INR <2 within the last 7 days prior to the ablation in patients receiving anticoagulants, and an INR <1.5 for patients not treated with anticoagulants.
* Platelets level >50 x 109/L within the last 7 days prior to the ablation.

Exclusion Criteria:

* Patients who decline or are unable to understand, provide or are unwilling to sign an informed consent form.
* Pregnant or nursing (lactating) women; women of childbearing potential and sexually active that are unwilling to use adequate contraception (such as oral contraceptives, intrauterine contraceptive device or barrier method with spermicide or surgical sterilization).
* Targeted tumor not clearly separated (i.e. located in the same liver segment as another tumor).
* Targeted tumor located in liver segments 1, 7 or 8.
* Targeted tumor >3 cm.
* Tumor that will be targeted >10 cm from the skin surface.
* Tumor not clearly visible with diagnostic ultrasound and MRI.
* Liver function score of Child-Pugh C.
* Liver volume reserve <40% as measured by CT Scan (54).
* Major surgical procedure, biopsy or significant traumatic injury <2 weeks prior to the procedure or has not recovered from side effects/complications of such procedure or trauma.
* Patient who has not recovered to grade 1 or better from any AEs (except alopecia, fatigue, nausea, vomiting) related to previous anti neoplastic therapies.
* BMI >30.
* Parkinson's disease.
* History of bleeding disorders (e.g. von Willebrand disease) or patients suspected to have a bleeding disorder.
* Not able to temporarily discontinue warfarin, clopidogrel or any other long-acting anticoagulants at least two weeks before the procedure.
* Initiation of any anticancer treatment during the screening period and during the follow-up study visits.
* Life expectancy to be less than 6 months.
* Unable or unwilling to complete all required screening and/or follow-up assessments.
* Patients under ongoing treatment with an investigational medication or medical device that conflicts with the study device.
* Patients for whom the investigator considers that the ablation is not in the patient's best interest.
* Patients with active alcohol or drug addiction or any other condition that, in the investigator's opinion, would interfere with their ability to comply with the study requirements.
* Patients with any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol.
* Patients with known sensitivity to iodine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Vidal Jove, MD, Principal Investigator — Mutua Terrassa , Barcelona, Spain
Locations (3):
- Spain (3):
  - Clinica Diagonal, Esplugues de Llobregat, Barcelona
  - Hospital universitario Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitario Vall d´Hebrón, Barcelona

REFERENCES:
- [Derived] Vidal-Jove J, Serres X, Vlaisavljevich E, Cannata J, Duryea A, Miller R, Merino X, Velat M, Kam Y, Bolduan R, Amaral J, Hall T, Xu Z, Lee FT Jr, Ziemlewicz TJ. First-in-man histotripsy of hepatic tumors: the THERESA trial, a feasibility study. Int J Hyperthermia. 2022;39(1):1115-1123. doi: 10.1080/02656736.2022.2112309. PMID 36002243

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Lesions
Period: Overall Study
Arm/Group | VORTX Rx Treatment
Started | 8; 11 Lesions
Completed | 5; 6 Lesions
Not Completed | 3; 5 Lesions

BASELINE CHARACTERISTICS:
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 8
Type of live tumors [Count of Participants; unit: Participants]
  Hepatocellular carcinoma | 1
  Liver metastasis | 7
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 25.1 [18.9 to 28.8]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0 - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. - Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
  Participants
    ECOG 0 | 2
    ECOG 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Acute Technical Performance of the VORTX Rx® Medical Device for the Ablation of Primary and Metastatic Liver Tumors
Description: Number of Lesions that were Successfully Ablated according to technical success definition established in the protocol.
Time Frame: 1-day post ablation
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 8
Number analyzed (lesions) | 11
lesions | 11

2. Secondary Outcome: Safety Profile of the VORTX Rx. Incidence of Adverse Events (Serious and Non-serious) That Are Probably or Definitely Device-related
Description: Number of Adverse Events (Serious and Non-serious) That Are Probably or Definitely Device-related
Time Frame: 2 months
Population: Although only 5 participants performed all protocol visits, adverse events from all patients were reported and analyzed.
  Any of the 55 AEs reported was device-related.
Measure: Number; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 8
Number analyzed (Adverse Events) | 55
Adverse Events | 0

3. Secondary Outcome: Local Tumor Progression
Description: Number of patients who have indicated local tumor progression in at least one visit (1 week, 1 month, 2 months) for each tumor ablated.
  The ablation zone will be assessed post-procedurally to evaluate local tumor progression by contrast-enhanced MRI imaging
Time Frame: 1 week, 1 month and 2 months post-procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 8
Participants
  Progression: YES | 2
  Progression: NO | 5
  Progression: No data | 1

4. Secondary Outcome: Involution of the Ablation Zone
Description: The involution of the ablation zone will be assessed post-procedurally by contrast-enhanced MRI imaging at 24h, 1 week, 1 month and 2 months
Time Frame: 24hours, 1 week, 1 month and 2 months, post-procedure.
Measure: Mean (Standard Deviation); unit: cubic centimeters
Units Other Than Participants: lesions
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 5
Number analyzed (lesions) | 6
cubic centimeters
  Ablation zone volume (cm3): 24 hours | 10.5500 (6.34405)
  Ablation zone volume (cm3): 1 week | 8.5000 (9.56682)
  Ablation zone volume (cm3): 1 month | 5.9383 (10.02174)
  Ablation zone volume (cm3): 2 months | 4.7683 (9.47795)

5. Secondary Outcome: Assessment of Liver panel_Part 1
Description: Liver panel will be evaluated on the basis of the change of aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase, gamma glutamyl transpeptidase (GGT) from baseline to evaluation visits 24 hours, 1 week and 1 and 2 months post procedure.
Time Frame: Screening, 24 hours, 1 week, 1 month and 2 months.
Population: Only 4 patients have these parameters determined in all study points (screening, 24h, 1 day, 1 month and 2 months post-ablation)
Measure: Mean (Standard Deviation); unit: U/L
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
U/L
  AST Screening | 60.7500 (33.83662)
  AST 24 hours | 183.5000 (80.71555)
  AST 1 week | 47.0000 (25.17936)
  AST 1 month | 40.7500 (10.68878)
  AST 2 months | 40.5000 (19.94158)
  ALT Screening | 44.0000 (22.13594)
  ALT 24 hours | 139.0000 (56.12486)
  ALT 1 week | 58.5000 (30.27100)
  ALT 1 month | 27.5000 (12.60952)
  ALT 2 months | 30.0000 (15.55635)
  GGT Screening | 127.2500 (105.05673)
  GGT 24 hours | 118.0000 (111.48692)
  GGT 1 week | 159.7500 (176.57364)
  GGT 1 month | 162.5000 (139.50986)
  GGT 2 months | 102.5000 (43.23964)
  Alkaline Phosphatase Screening | 156.5000 (139.89639)
  Alkaline Phosphatase 24 hours | 127.2500 (67.14847)
  Alkaline Phosphatase 1 week | 165.0000 (88.67168)
  Alkaline Phosphatase 1 month | 146.7500 (66.33941)
  Alkaline Phosphatase 2 months | 130.2500 (74.44629)

6. Secondary Outcome: Assessment of Liver Panel_Part 2
Description: Liver panel will be evaluated on the basis of the change of albumin from baseline to evaluation visits 24 hours, 1 week and 1 and 2 months post procedure.
Time Frame: 24 hours, 1 week and 1 month and 2 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/L
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
g/L
  Albumin Screening | 40.0250 (2.88603)
  Albumin 24 hours | 34.7500 (1.13284)
  Albumin 1 week | 37.5250 (1.95683)
  Albumin 1 month | 39.3750 (0.63966)
  Albumin 2 months | 40.1750 (1.65806)

7. Secondary Outcome: Assessment of Liver Panel_Part 3
Description: Liver panel will be evaluated on the basis of the change of bilirubin from baseline to evaluation visits 24 hours, 1 week and 1 and 2 months post procedure
Time Frame: 24 hours, 1 week and 1month and 2 months
Measure: Mean (Standard Deviation); unit: mg/dL
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
mg/dL
  Total Bilirrubin Screening | 0.7525 (0.42578)
  Total Bilirrubin 24 hours | 0.6425 (0.20549)
  Total Bilirrubin 1 week | 0.7600 (0.32934)
  Total Bilirrubin 1 month | 0.5250 (0.11561)
  Total Bilirrubin 2 months | 0.7050 (0.31268)

8. Secondary Outcome: Assessment of Liver Panel_part 4
Description: Liver panel will be evaluated on the basis of the change of prothrombin time (PT) from baseline to evaluation visits 24 hours, 1 week and 1 and 2 months post procedure
Time Frame: 24 hours, 1 week and 1month and 2 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of activity
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
percentage of activity
  Prothrombin time Screening | 95.2500 (5.50000)
  Prothrombin time 24 hours | 92.5000 (9.94987)
  Prothrombin time 1 week | 92.7500 (8.38153)
  Prothrombin time 1 month | 98.7500 (2.50000)
  Prothrombin time 2 months | 91.2500 (17.50000)

9. Secondary Outcome: Assessment of Liver Panel_Part 5
Description: Liver panel will be evaluated on the basis of the change of International normalized ratio (INR = A system established by the World Health Organization (WHO) and the International Committee on Thrombosis and Hemostasis for reporting the results of blood coagulation (clotting) tests) from baseline to evaluation visits 24 hours, 1 week and 1 and 2 months post procedure.
  The INR is derived from prothrombin time (PT) which is calculated as a ratio of the patient's PT to a control PT standardized for the potency of the thromboplastin reagent developed by the World Health Organization (WHO) using the following formula: INR = Patient PT ÷ Control PT.
  Normal values for INR: 0.9-1.3.
Time Frame: 24 hours, 1 week and 1 month and 2 months
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
ratio
  INR Screening | 1.0500 (0.5774)
  INR 24 hours | 1.0750 (0.09574)
  INR 1 week | 1.0500 (0.05774)
  INR 1 month | 1.0250 (0.05000)
  INR 2 months | 1.0750 (0.15000)

10. Secondary Outcome: Immunologic Assessment_Part 1
Description: Immunological response of ablation will be evaluated on the basis of immune tests conducted and tumor biomarker assessments (including, but not limited to, immune tests: CD3+, CD4+, CD8+, CD45+, CD16+, CD56+ and CD19+ from Baseline/Screening to 1-day post ablation, 1 week and 1 and 2 months post procedureprocedure.
Time Frame: Baseline/Screening, 1-day post ablation, 1 week and 1 and 2 months post procedure
Measure: Mean (Standard Deviation); unit: cells/uL
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
cells/uL
  CD3+ (T cells) Screening | 801.7500 (374.33708)
  CD3+ (T cells) 24 hours | 618.2500 (365.48814)
  CD3+ (T cells) 1 week | 713.7500 (234.09596)
  CD3+ (T cells) 1 month | 587.7500 (253.11575)
  CD3+ (T cells) 2 months | 632.0000 (150.53017)
  CD4+ (T helper cells) Screening | 469.2500 (146.20619)
  CD4+ (T helper cells) 24 hours | 374.7500 (128.99709)
  CD4+ (T helper cells) 1 week | 445.2500 (121.94637)
  CD4+ (T helper cells) 1 month | 357.0000 (159.34240)
  CD4+ (T helper cells) 2 months | 382.2500 (77.24150)
  CD8+ (T suppressor/cytotoxic cells) Screening | 262.7500 (223.82638)
  CD8+ (T suppressor/cytotoxic cells) 24 hours | 220.5000 (204.31593)
  CD8+ (T suppressor/cytotoxic cells) 1 week | 230.5000 (139.01679)
  CD8+ (T suppressor/cytotoxic cells) 1 month | 186.7500 (136.19196)
  CD8+ (T suppressor/cytotoxic cells) 2 months | 177.2500 (85.47660)
  CD45+ (leucocyte common antigen) Screening | 1054.1425 (384.46746)
  CD45+ (leucocyte common antigen) 24 hours | 843.0350 (349.94733)
  CD45+ (leucocyte common antigen) 1 week | 938.3700 (251.60549)
  CD45+ (leucocyte common antigen) 1 month | 788.4275 (257.71702)
  CD45+ (leucocyte common antigen) 2 months | 831.2675 (194.76464)
  CD16+ Screening | 134.3000 (69.78811)
  CD16+ 24 hours | 78.4750 (50.40353)
  CD16+ 1 week | 116.1750 (65.72460)
  CD16+ 1 month | 109.7500 (53.11230)
  CD16+ 2 months | 100.5000 (47.59202)
  CD56+ (NKT cells) Screening | 85.4500 (85.14507)
  CD56+ (NKT cells) 24 hours | 56.5000 (61.00213)
  CD56+ (NKT cells) 1 week | 73.9500 (69.58934)
  CD56+ (NKT cells) 1 month | 63.2500 (68.07533)
  CD56+ (NKT cells) 2 months | 60.7500 (50.12900)
  CD19+ (B-lymphocyte antigen) Screening | 85.0000 (58.66856)
  CD19+ (B-lymphocyte antigen) 24 hours | 83.5000 (58.31238)
  CD19+ (B-lymphocyte antigen) 1 week | 86.5000 (53.10053)
  CD19+ (B-lymphocyte antigen) 1 month | 70.0000 (50.51732)
  CD19+ (B-lymphocyte antigen) 2 months | 87.0000 (51.71718)

11. Secondary Outcome: Immunologic Assessment_Part 2
Description: Immunological response of ablation will be evaluated on the basis of immune tests conducted and tumor biomarker assessments: C-reactive protein [CRP], from baseline to evaluation visits 1 day, 1 week and 1 and 2 months post procedure.
Time Frame: Screening, 24 hours, 1 week and 1 and 2 months post procedure.
Measure: Mean (Standard Deviation); unit: mg/L
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
mg/L
  C reactive protein Screening | 5.9750 (5.67355)
  C reactive protein 24 hours | 6.0250 (7.06323)
  C reactive protein 1 week | 30.8250 (53.05735)
  C reactive protein 1 month | 4.7750 (3.57713)
  C reactive protein 2 months | 11.9500 (8.85795)

12. Secondary Outcome: Immunologic Assessment_Part 3
Description: Immunological response of ablation will be evaluated on the basis of immune tests conducted and tumor biomarker assessments (including, but not limited to, immune tests): complement C3 and C4, immunoglobulins [IgG, IgM, IgA] from baseline to evaluation visits 1 day, 1 week and 1 and 2 months post procedure.
Time Frame: Screening, 24 hours post ablation, 1 week and 1 and 2 months post procedure.
Measure: Mean (Standard Deviation); unit: mg/dL
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
mg/dL
  Complement C3 Screening | 144.0000 (53.61592)
  Complement C3 24 hours | 123.2000 (25.76354)
  Complement C3 1 week | 150.5000 (22.75229)
  Complement C3 1 month | 143.9000 (44.60239)
  Complement C3 2 months | 134.7500 (26.88711)
  Complement C4 Screening | 30.7750 (20.29949)
  Complement C4 24 hours | 23.7750 (6.58401)
  Complement C4 1 week | 29.8250 (9.00717)
  Complement C4 1 month | 26.9500 (11.01348)
  Complement C4 2 months | 28.0750 (14.47236)
  IgG Screening | 867.2500 (326.38359)
  IgG 24 hours | 792.9000 (354.83048)
  IgG 1 week | 856.0000 (335.22430)
  IgG 1 month | 916.7500 (338.63784)
  IgG 2 months | 899.0000 (334.19655)
  IgM Screening | 132.6250 (59.75139)
  IgM 24 hours | 120.9000 (51.44745)
  IgM 1 week | 132.3500 (45.62846)
  IgM 1 month | 140.7500 (43.69115)
  IgM 2 months | 141.2500 (52.94075)
  IgA Screening | 147.5000 (133.49871)
  IgA 24 hours | 130.0000 (119.05766)
  IgA 1 week | 142.8000 (131.15955)
  IgA 1 month | 145.9500 (116.11530)
  IgA 2 months | 129.3750 (84.51147)

13. Secondary Outcome: Immunologic Assessment_Part 4
Description: Immunological response of ablation will be evaluated on the basis of immune tests conducted and tumor biomarker assessments (including, but not limited to, immune tests: complement CH50, alfa-fetoprotein [AFP], Cancer Antigens CA15-3 [Breast Cancer] and CA 19-9 [Pancreatic Cancer]) from baseline to evaluation visits 1 day, 1 week and 1 and 2 months post procedure.
Time Frame: Screening, 24 hours post ablation, 1 week and 1 and 2 months post procedure.
Measure: Mean (Standard Deviation); unit: U/ml
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
U/ml
  Complement CH50 Screening | 72.7500 (26.87471)
  Complement CH50 24 hours | 61.5000 (37.59876)
  Complement CH50 1 week | 61.0000 (34.02940)
  Complement CH50 1 month | 52.2500 (24.18505)
  Complement CH50 2 months | 60.2500 (36.59121)
  AFP Screening | 544.8050 (1084.79682)
  AFP 24 hours | 417.8550 (831.43014)
  AFP 1 week | 502.2350 (999.84372)
  AFP 1 month | 264.1675 (523.22173)
  AFP 2 months | 224.5900 (441.61247)
  CA 15-3 (breast cancer) Screening | 15.8500 (9.02940)
  CA 15-3 (breast cancer) 24 hours | 14.0000 (6.66433)
  CA 15-3 (breast cancer) 1 week | 14.3750 (7.20804)
  CA 15-3 (breast cancer) 1 month | 16.2250 (9.31786)
  CA 15-3 (breast cancer) 2months | 15.4250 (7.08396)
  CA 19-9 (pancreatic cancer) Screening | 167.8175 (300.24702)
  CA 19-9 (pancreatic cancer) 24 hours | 174.8450 (312.86710)
  CA 19-9 (pancreatic cancer) 1 week | 169.1675 (290.56204)
  CA 19-9 (pancreatic cancer) 1 month | 168.1200 (285.77017)
  CA 19-9 (pancreatic cancer) 2 months | 256.9525 (475.14915)

14. Secondary Outcome: Immunologic Assessment_Part 5
Description: Immunological response of ablation will be evaluated on the basis of immune tests conducted and tumor biomarker assessments (including, but not limited to, immune tests): interleukin-6 [IL-6] from baseline to evaluation visits 1 day, 1 week and 1 and 2 months post procedure.
Time Frame: Screening, 24 hours post ablation, 1 week and 1 and 2 months post procedure.
Measure: Mean (Standard Deviation); unit: pg/dl
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
pg/dl
  Interleukin-6 Screening | 4.2225 (2.88648)
  Interleukin-6 24 hours | 3.4575 (1.97481)
  Interleukin-6 1 week | 14.7850 (14.05719)
  Interleukin-6 1 month | 3.8750 (2.37905)
  Interleukin-6 2 months | 5.8125 (2.84372)

15. Secondary Outcome: Immunologic Assessment_Part 6
Description: Immunological response of ablation will be evaluated on the basis of immune tests conducted and tumor biomarker assessments (including, but not limited to, immune tests): carcinoembryonic antigen [CEA] from baseline to evaluation visits 1 day, 1 week and 1 and 2 months post procedure.
Time Frame: Screening, 24 hours post ablation, 1 week and 1 and 2 months post procedure.
Measure: Mean (Standard Deviation); unit: ng/ml
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
ng/ml
  CEA Screening | 46.9300 (50.75086)
  CEA 24 hours | 50.4200 (55.16530)
  CEA 1 week | 37.7925 (45.10227)
  CEA 1 month | 44.6150 (64.11322)
  CEA 2 months | 54.0225 (97.45371)

16. Secondary Outcome: Assesment of Quality of Life by Using Patient Questtionaires EORTC QLQ-C30. (European Organization for Research and Treatment of Cancer)
Description: The EORTC QLQ-C30 is a 30-item generic health-related QoL instrument designed to assess cancer patients' physical, psychological and social functioning. It is composed of 9 multi-item scales (5 functional scales [physical, role, cognitive, emotional, and social], a global QoL scale [GQoL], and 3 symptom scales [fatigue, pain, and nausea and vomiting]), 5 single-item symptom scales assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhea), and an item on the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0-100. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/QoL represents a high QoL. However, a high score for a symptom scale/item represents a high level of symptomatology/problems.
Time Frame: Screening, 1 and 2 months post procedure.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 4
Number analyzed (ablation procedures) | 4
score on a scale
  Global health status/QoL Screening | 70.8333 (15.95712)
  Global health status/QoL 1 month | 58.3333 (28.05418)
  Global health status/QoL 2 months | 70.8333 (25.00000)
  Physical functioning Screening | 81.6667 (12.61980)
  Physical functioning 1 month | 83.3333 (13.87777)
  Physical functioning 2 months | 81.6667 (18.35857)
  Role functioning screening | 87.5000 (15.95712)
  Role functioning 1 month | 70.8333 (28.46375)
  Role functioning 2 months | 83.3333 (13.60828)
  Emotional functioning Screening | 87.5000 (8.33333)
  Emotional functioning 1 month | 87.5000 (19.83730)
  Emotional functioning 2 months | 83.3333 (18.00206)
  Cognitive functioning Screening | 79.1667 (20.97176)
  Cognitive functioning 1 month | 75.0000 (21.51657)
  Cognitive functioning 2 months | 79.1667 (31.54949)
  Social functioning Screening | 95.8333 (8.33333)
  Social functioning 1 month | 83.3333 (13.60828)
  Social functioning 2 months | 95.8333 (8.33333)
  Fatigue Screening | 30.5556 (13.98117)
  Fatigue 1 month | 41.6667 (27.77778)
  Fatigue 2 months | 25.0000 (24.63729)
  Nausea and vomiting Screening | 0 (0)
  Nausea and vomiting 1 month | 0 (0)
  Nausea and vomiting 1 months | 0 (0)
  Pain Screening | 16.6667 (23.57023)
  Pain 1 month | 20.8333 (31.54949)
  Pain 2 months | 41.6667 (34.69443)
  Dyspnea Screening | 0 (0)
  Dyspnea 1 month | 0 (0)
  Dyspnea 2 months | 0 (0)
  Insomnia Screening | 41.6667 (41.94352)
  Insomnia 1 month | 33.3333 (47.14045)
  Insomnia 2 months | 25.0000 (31.91424)
  Appetite loss Screening | 25.0000 (50.00000)
  Appetite loss 1 month | 50.0000 (43.03315)
  Appetite loss 2 months | 8.3333 (16.66667)
  Constipation Screening | 8.3333 (16.66667)
  Constipation 1 month | 0 (0)
  Constipation 2 months | 0 (0)
  Diarrhea Screening | 33.3333 (47.14045)
  Diarrhea 1 month | 16.6667 (19.24501)
  Diarrhea 2 months | 16.6667 (19.24501)
  Financial difficulties Screening | 16.6667 (19.24501)
  Financial difficulties 1 month | 8.3333 (16.66667)
  Financial difficulties 2 months | 8.3333 (16.66667)

17. Secondary Outcome: Pain Assessment by VAS Scale
Description: Perform pain assessment by a 100 mm visual analog scale (VAS) where 0 is "no pain" and 100 is "the maximum pain possible" at 1-day and 1-week post-procedure.
Time Frame: 1-day post ablation and 1 week post procedure.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: ablation procedures
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 7
Number analyzed (ablation procedures) | 7
score on a scale
  VAS score: 24 hours | 4.3 (7.9)
  VAS score: 1 week | 25.0 (18.9)

18. Secondary Outcome: Analgesic Requirements After the Ablation Procedure
Description: Evaluate analgesic treatment prescription in the 24-hour period post-procedure and during the one week period post-procedure.
Time Frame: in the 24-hour period post-procedure and during the one week period post-procedure
Population: Number of patients with at least one drug due to Post-procedure pain (concomitant medication form).
Measure: Count of Participants; unit: Participants
Arm/Group | VORTX Rx Treatment
Number analyzed (Participants) | 8
Participants
  At least one drug due to post-procedure pain: YES | 5
  At least one drug due to post-procedure pain: NO | 3

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | VORTX Rx Treatment
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VORTX Rx Treatment (N=8)
FEVER (General disorders) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VORTX Rx Treatment (N=8)
Transaminase elevation (Hepatobiliary disorders) | 1
Abdominal discomfort (General disorders) | 1
Abdominal pain (General disorders) | 1
Adverse reaction to analeptics and opioid receptor antagonists (Nervous system disorders) | 1
Alkaline phosphatase increase (Hepatobiliary disorders) | 1
ALT increase (Hepatobiliary disorders) | 4
Anemia (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Appetite increase (Metabolism and nutrition disorders) | 1
Ascites (Hepatobiliary disorders) | 1
AST increase (Hepatobiliary disorders) | 4
Chest punctures (Respiratory, thoracic and mediastinal disorders) | 1
Choluria (Renal and urinary disorders) | 1
Coccyx pain (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Desquamative lesions (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
General pain (General disorders) | 1
GGT increase (Hepatobiliary disorders) | 2
Itchy skin (Skin and subcutaneous tissue disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Left leg pain (Musculoskeletal and connective tissue disorders) | 1
Lipotomy (Nervous system disorders) | 1
Malleolar edema with fovea (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Occasional fever (General disorders) | 1
Pain in right shoulder (Musculoskeletal and connective tissue disorders) | 1
Pain in right side (Musculoskeletal and connective tissue disorders) | 1
Right basal pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Sciatic pain (Nervous system disorders) | 3
Swollen ankles (Vascular disorders) | 1
Tingling in feet and hands (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results or conclusions of this study will be reported at scientific congresses and published in scientific journals. The investigator agrees to maintain this information in strict confidence, and will not use it for any other purpose without the written authorization of the sponsor.

DOCUMENTS (3):
  • Study Protocol (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT03741088/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03741088/SAP_001.pdf
  • Informed Consent Form (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT03741088/ICF_002.pdf